CLINICAL TRIAL: NCT02354703
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Pharmacogenetic Study of Ondansetron in Alcohol Use Disorder
Brief Title: Pharmacogenetic Study of Ondansetron in Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Gorelick, MD, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP00061575
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Use Disorder
Keywords: alcoholism, treatment, serotonin transporter
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design: treatment intervention (active, placebo) x genotype (responsive, non-responsive)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: treatment assignment and genotype classification known only to research pharmacist and study biostatistician who performed randomization.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ondansetron-responsive genotype (Experimental): ondansetron-0.33 mg bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and carrying one of the following genotypes:
  if European ancestry:
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  HTR3A gene:
  rs1150226:AG; or rs1176713:GG
  HTR3B gene:
  rs17619942:AC
  If African ancestry:
  HTR3B gene:
  rs176744: CC or CA
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  Interventions: Drug: Ondansetron
- ondansetron--non-responsive genotype (Experimental): ondansetron-0.33 mg bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and NOT carrying any of the responsive genotypes
  Interventions: Drug: Ondansetron
- placebo--responsive genotype (Placebo Comparator): placebo bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and carrying one of the following genotypes:
  if European ancestry:
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  HTR3A gene:
  rs1150226:AG; or rs1176713:GG
  HTR3B gene:
  rs17619942:AC
  If African ancestry:
  HTR3B gene:
  rs176744: CC or CA
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  Interventions: Drug: Placebo
- placebo--non-responsive genotype (Placebo Comparator): placebo bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and NOT carrying any of the responsive genotypes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Ondansetron (0.33 mg) bid+ BBCET counseling
  Arms: ondansetron--non-responsive genotype; ondansetron-responsive genotype
Drug: Placebo — Placebo + BBCET counseling
  Arms: placebo--non-responsive genotype; placebo--responsive genotype

SUMMARY:
The primary study objective is to determine the efficacy of ondansetron (0.33 mg twice daily) administered orally for a period of 16 weeks in reducing risky drinking among currently drinking subjects with alcohol use disorder who have selected genotypes at the serotonin transporter and receptor genes. The secondary objective is to assess the safety and tolerability of ondansetron in subjects with alcohol use disorder who have selected genotypes at the serotonin transporter and receptor genes.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a heterogeneous and chronic relapsing disorder that includes both acute (binge drinking) and chronic (frequent heavy drinking) dimensions. Perhaps because of this heterogeneity, the therapeutic effect size of the approved medicines for the treatment of AUD has been small. In an effort to overcome the heterogeneity of response to a particular medication, recent studies have instituted a personalized approach to therapy. Major breakthroughs in pharmacogenetics have made it possible to identify discrete subgroups of the AUD population according to genetic profiles in order to target the subjects who are most likely to respond to treatment with a particular agent. In addition, genetic variation contributing to the risk of alcohol dependence may be differentially associated with treatment response Thus a successful personalized medicinal approach should ensure that targeted subgroups achieve an optimal treatment response with high predictability. Such an approach holds the potential to identify not only robust responders to treatment but also those who might have minimal or modest adverse effects from the putative therapeutic medication. From a practical clinical standpoint, a personalized medicine approach starts with a genetic screen to identify the "right" subject, who can then be treated with the appropriate medication, with a high probability of a positive treatment outcome and, therefore, a substantial impact on public health.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who have given written informed consent
* Aged 18 to 70
* The subject has a breath alcohol concentration (BrAC) = 0.00% at the screening visit and < or = 0.02% at all visits after the screening visit
* Diagnosis of alcohol use disorder (AUD) using Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria
* Able to provide Time-Line Follow-Back (TLFB) alcohol consumption information for the 90-day period prior to the Screen Visit.
* During the 4 weeks preceding the Baseline Visit, the subject reports:

  * ≥6 Heavy Drinking Days (HDDs) - defined as a day with alcohol consumption of ≥5 standard drinks (i.e., 12 g of ethanol) for men, and ≥ 4 standard drinks for women
  * ≤14 consecutive abstinent days
  * Total alcohol consumption of an average of ≥21 standard drinks/week for men and ≥14 standard drinks/week for women in past 28 days and have met these criteria during the 7 days prior to randomization
* An expressed wish to reduce or stop drinking
* Willingness to participate in behavioral and medicinal treatments for AUD
* Stable residence in the 28 days prior to the Baseline Visit and no plans to move in the next 9 months. A stable residence is a domicile in which an individual can operate as if it were his or her own homestead and does not include shelters or halfway houses.
* Provides contact information for 1 or 2 "locators" who can be used to contact the subject
* Able to read and understand English and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments. This will be assessed with the Slosson Oral Reading Test-Revised, on which the subject must demonstrate at least a 6th grade reading level.
* If the subject is a woman of child-bearing age, she must:
* Agree not to try to become pregnant during the study, and use adequate contraception (defined as oral/ systemic contraception, intrauterine device, diaphragm in combination with spermicide, or condom for male partner in combination with spermicide) or
* Be postmenopausal, (i.e., have had her last natural menstruation at least 24 months prior to baseline) or
* Have had a hysterectomy or been surgically sterilized prior to the Baseline Visit, or
* Plan not to be sexually active vaginally with men during the entire duration of the trial.

Exclusion Criteria:

* A subject presenting with any of the following at the Baseline Visit will be excluded from the study:

  * The subject has fewer than 6 heavy drinking days (HDD) (defined as ≥5 standard drinks for men and ≥4 or greater standard drinks for women) in the 4 weeks preceding the Baseline Visit.
  * The subject has greater than 14 consecutive abstinent days in the 4 weeks preceding the Baseline Visit.
  * The subject has a Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar), Revised, score ≥10
  * The subject has a current diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder, or a non-psychotic diagnosis such as major depressive disorder, post-traumatic stress disorder, panic disorder, eating disorder, or substance use disorder (except alcohol, tobacco, or cannabis) that is judged by the PI or designee as exclusionary.
  * Current or recent (within 4 weeks prior to Baseline Visit) treatment with antipsychotics or any medication likely to interact with ondansetron to produce an adverse effect, as judged by a study physician.
  * Treatment with any investigational medicinal product within 30 days or 5 half-lives (whichever is longer) prior to Randomization.
  * Currently participating or has recently (4 weeks prior to Randomization) participated in a treatment program for alcohol use disorders.
  * Mini-International Neuropsychiatric Interview (MINI) 6.0 Suicide Risk Assessment module B will be used to assess subjects' risk of suicide. A score of > or = 9 will be evaluated by the PI or designee to determine eligibility. Subjects who are deemed by the PI or designee to be at risk of suicide will be excluded.
  * Clinically significant, unstable physical illness (e.g., hematologic, hepatic or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance), as judged by the PI or designee to be exclusionary
  * Clinically significant abnormal vital signs, as judged by the PI or designee
  * Clinically significant abnormal 12-lead ECG at the Screen Visit, clinically significant cardiovascular disease requiring regular or intensive clinical monitoring, a current history of arrhythmias, or a current or past history of clinically significant QT prolongation, including: QTcF > 450 ms (average of 3 12-lead measurements)

    * Serum potassium, magnesium or calcium levels outside the central laboratory's reference range that are deemed clinically significant by the PI or designee.
    * Taking medications (within the last 7 days prior to the Baseline Visit) that have the potential to prolong the QT interval, as judged by a study physician, or may require such medications during the course of the study. For patients taking these medications, a study physician will evaluate the potential for ondansetron to interact with the medication to produce a clinically significant risk for the participant.
    * Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia or indwelling cardiac pacemaker
    * Complete left bundle branch block
    * History of Long QT Syndrome or a first-degree biological family member with this condition
  * Evidence of hepatic failure and/or ascites, prolonged prothrombin time (International Normalized Ratio [INR] > or = 1.7), bilirubin >10% above the upper limit of the central lab's normal range and/or esophageal variceal disease
  * Active hepatitis and/or serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) or lactate dehydrogenase (LDH) > 3x the upper limit of normal
  * Treatment, either current or within 28 days prior to Randomization, with any medications having a potential effect on alcohol consumption and related behaviors or mood. These include opioid antagonists (e.g., naltrexone, Vivitrol®, Selincro®), glutamate antagonists (e.g., acamprosate), anticonvulsants (e.g., topiramate, gabapentin), serotonin reuptake inhibitors (e.g., fluoxetine), serotonin antagonists (e.g., buspirone), other antidepressants (e.g., tricyclic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g., haloperidol), and disulfiram (Antabuse®)
  * At the Screen Visit, the subject's urine contains opiates, cocaine, amphetamines, barbiturates, or benzodiazepines that cannot be explained by appropriate use of prescribed medication
  * History of severe or life-threatening adverse reactions to ondansetron
  * Female subjects of childbearing potential who have a positive pregnancy test at Baseline Visit or are pregnant, breast feeding, not adhering to an acceptable form of contraception at screening or any time during the study, or unwilling to maintain an acceptable form of contraception throughout the study
  * Prior to Randomization, the subject is compelled to participate in an alcohol treatment program to maintain his/her liberty
  * As of Screen Visit, the subject is sharing a household with a subject randomized to any investigational trial of ondansetron
  * Any other condition or therapy that, in the investigator's opinion, may pose a risk to the subject, prevent the subject from completing the required study procedures or interfere with the study objectives • Less than 75% European ancestry proportions or African-American ancestry proportions

    * Body weight greater than or equal to 110 kg (242 lb)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Gorelick, MD, PhD, Principal Investigator — University of Maryland, Baltimore; Henry R Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - MPRC, Baltimore, Maryland
  - University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania
  - Philadelphia VAMC, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from August, 2015 through December 2019 in the Philadelphia, PA and Baltimore, MD metropolitan areas using print, broadcast, and internet advertising, referral from local clinics, and search of medical records for potential participants.
Pre-assignment Details: 293 participants were enrolled, which allowed them to be screened for study eligibility. 115 participants meet eligibility criteria and were scheduled for randomization. 6 participants did not remain eligible at baseline visit and 14 participants did not appear at the baseline visit, resulting in 95 participants randomized and starting treatment.
Groups:
- Ondansetron-responsive Genotype: ondansetron-0.33 mg bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and carrying one of the following genotypes:
  if European ancestry:
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  HTR3A gene:
  rs1150226:AG; or rs1176713:GG
  HTR3B gene:
  rs17619942:AC
  If African ancestry:
  HTR3B gene:
  rs176744: CC or CA
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  Ondansetron: Ondansetron (0.33 mg) bid+ BBCET counseling
- Placebo--responsive Genotype: placebo bid + Brief Behavioral Compliance Enhancement Treatment (BBCET) for 16 weeks and carrying one of the following genotypes:
  if European ancestry:
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  HTR3A gene:
  rs1150226:AG; or rs1176713:GG
  HTR3B gene:
  rs17619942:AC
  If African ancestry:
  HTR3B gene:
  rs176744: CC or CA
  SLC6A4 gene:
  5-HTTLPR:LL, or rs25531:AA, or 5-HTTLPR + rs25531 (LALA genotype) or rs1042173:TT
  Placebo: Placebo + BBCET counseling
Period: Overall Study
Arm/Group | Ondansetron--non-responsive Genotype | Ondansetron-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype
Started | 12 | 34 | 39 | 10
Completed | 9 | 26 | 28 | 7
Not Completed | 3 | 8 | 11 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 7 | 9 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron--non-responsive Genotype | Ondansetron-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype | Total
Number analyzed (Participants) | 12 | 34 | 39 | 10 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.58 (6.96) | 52.29 (10.59) | 49.33 (12.07) | 53.10 (14.04) | 51.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 10 | 4 | 26
  Male | 8 | 26 | 29 | 6 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 11 | 34 | 37 | 10 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 17 | 16 | 1 | 35
  White | 11 | 17 | 23 | 9 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 34 | 39 | 10 | 95
marital status [Count of Participants; unit: Participants] — number of married participants
  Participants | 5 | 14 | 26 | 5 | 50
employment status [Count of Participants; unit: Participants] — number of employed (full- or part-time) participants
  Participants | 8 | 31 | 27 | 8 | 74
education level [Mean (Standard Deviation); unit: years] | 15.06 (2.64) | 15.82 (3.79) | 15.33 (3.09) | 17.80 (1.55) | 15.7 (3.2)
lifetime major depressive disorder [Count of Participants; unit: Participants] | 1 | 4 | 5 | 2 | 12
lifetime anxiety disorder [Count of Participants; unit: Participants] | 0 | 7 | 3 | 0 | 10
Beck Depression Inventory (BDI) score [Mean (Standard Deviation); unit: units on a scale] — Total score on the Beck Depression Inventory (BDI), a 21-item self-report measure of depressive symptoms. Each item is a 0-3 LIkert scale. Total score ranges from 0 to 63, with higher scores indicating greater depression.
  units on a scale | 4.08 (4.12) | 6.53 (5.81) | 5.22 (5.13) | 2.33 (2.55) | 5.2 (5.2)
Short Index of Problems (SIP) [Mean (Standard Deviation); unit: units on at scale] — Total score on the Short Index of Problems (SIP), 15-item self-report instrument which measures adverse consequences of drinking. Each item is a 0-3 Likert scale. Total score ranges from 0 to 45, with higher scores indicating more severe alcohol-related problems.
  units on at scale | 14.33 (11.88) | 14.29 (9.68) | 12.51 (9.13) | 12.30 (6.11) | 13.4 (9.4)
drinks per drinking day (DPDD) [Mean (Standard Deviation); unit: drinks per drinking day] — self-reported number of standard drinks of alcohol (14 g alcohol) consumed per drinking day
  drinks per drinking day | 5.80 (2.50) | 6.77 (2.90) | 6.32 (2.69) | 6.56 (3.74) | 6.4 (2.8)
percent drinking days (PDD) [Mean (Standard Deviation); unit: percent of days with alcohol drinking] — self-reported percent of days on which the participant drank alcohol
  percent of days with alcohol drinking | 85.0 (20.49) | 86.73 (21.39) | 87.29 (16.54) | 88.0 (15.45) | 86.9 (18.5)
percent heavy drinking days (PHDD) [Mean (Standard Deviation); unit: percent of heavy drinking days] — self-reported percent of drinking days on which at least 5 standard drinks (14 g alcohol) for men or at least 4 standard drinks for women were consumed
  percent of heavy drinking days | 75.92 (24.79) | 75.72 (26.34) | 70.84 (25.7) | 78.56 (22.46) | 74.0 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: self-reported number of standard drinks of alcohol (14 g alcohol) consumed per drinking day
Time Frame: 16-week treatment period
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Ondansetron-responsive Genotype | Ondansetron--non-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype
Number analyzed (Participants) | 34 | 12 | 39 | 10
drinks per drinking day | 3.70 (2.44) | 3.60 (2.20) | 3.37 (2.35) | 3.99 (3.81)
Statistical Analysis 1: Comparison: Ondansetron-responsive Genotype vs Ondansetron--non-responsive Genotype vs Placebo--responsive Genotype vs Placebo--non-responsive Genotype; Test type: Superiority; p = 0.94, Kruskal-Wallis — a priori significance P<0.05; adjusted for baseline value

2. Secondary Outcome: Percent Drinking Days
Description: self-reported percentage of days on which the participant drank alcohol
Time Frame: 16-week treatment period
Measure: Mean (Standard Deviation); unit: percentage of drinking days
Arm/Group | Ondansetron--non-responsive Genotype | Ondansetron-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype
Number analyzed (Participants) | 12 | 34 | 39 | 10
percentage of drinking days | 71.92 (15.08) | 67.51 (26.33) | 68.00 (27.09) | 66.84 (34.39)
Statistical Analysis 1: Comparison: Ondansetron--non-responsive Genotype vs Ondansetron-responsive Genotype vs Placebo--responsive Genotype vs Placebo--non-responsive Genotype; Test type: Superiority; p = 1.00, Chi-squared — a priori significance is P<0.05; adjusted for baseline value

3. Secondary Outcome: Percent Heavy Drinking Days
Description: self-reported percentage of days with heavy drinking (at least 5 drinks/day for men, at least 4 drinks/day for women)
Time Frame: 16-week treatment period
Measure: Mean (Standard Deviation); unit: percentage of days with heavy drinking
Arm/Group | Ondansetron--non-responsive Genotype | Ondansetron-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype
Number analyzed (Participants) | 12 | 34 | 39 | 10
percentage of days with heavy drinking | 32.93 (23.59) | 40.49 (32.08) | 31.96 (27.27) | 35.13 (35.04)
Statistical Analysis 1: Comparison: Ondansetron--non-responsive Genotype vs Ondansetron-responsive Genotype vs Placebo--responsive Genotype vs Placebo--non-responsive Genotype; Test type: Superiority; p = 0.73, Kruskal-Wallis — a priori threshold is P<0.05; adjusted for baseline value

ADVERSE EVENTS:
Time Frame: 16-week treatment period
Description: Adverse events assessed by participant self-report. Many events were assessed without regard to a specific Adverse Event Term.
Arm/Group | Ondansetron--non-responsive Genotype | Ondansetron-responsive Genotype | Placebo--responsive Genotype | Placebo--non-responsive Genotype
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/34 | 0/39 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/34 | 1/39 | 0/10
Other Adverse Events (participants affected / at risk) | 10/12 | 30/34 | 34/39 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron--non-responsive Genotype (N=12) | Ondansetron-responsive Genotype (N=34) | Placebo--responsive Genotype (N=39) | Placebo--non-responsive Genotype (N=10)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not study-related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ondansetron--non-responsive Genotype (N=12) | Ondansetron-responsive Genotype (N=34) | Placebo--responsive Genotype (N=39) | Placebo--non-responsive Genotype (N=10)
nervous system (Nervous system disorders) | 3 | 12 | 13 | 3 — all adverse events affecting nervous system
gastrointestinal (Gastrointestinal disorders) | 3 | 10 | 12 | 2
infections (Infections and infestations) | 5 | 7/14 | 12 | 3
musculoskeletal & connective tissue (Musculoskeletal and connective tissue disorders) | 4 | 6 | 7 | 4
skin & subcutaneous tissue (Skin and subcutaneous tissue disorders) | 2 | 2 | 13 | 1
psychiatric (Psychiatric disorders) | 1 | 8 | 4 | 3
general disorders (General disorders) | 2 | 5 | 4 | 3
injury, poisoning, procedural (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 1
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
immune (Immune system disorders) | 0 | 4 | 1 | 0
eye (Eye disorders) | 0 | 0 | 3 | 1
blood & lymphatic (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
metabolism & nutrition (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
reproductive & breast (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
ear (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
renal & urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The pre-specified enrollment target of 256 participants starting treatment was calculated to detect a difference in change in drinks per drinking day between ondansetron and placebo groups at an effect size of 0.59 with a power of 0.84. The achieved enrollment of 95 participants was substantially below this pre-specified target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02354703/Prot_SAP_000.pdf